CLINICAL TRIAL: NCT04356105
Title: Minimal Stimulation in a Combined Letrozole Antagonist Protocol Versus Microflare Protocol in Poor Responders Undergoing Invitrofertilization/ Intracytoplasmic Sperm Injection; Randomized Parallel Study
Brief Title: Protocols of IVF/ICSI in Poor Responders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmin Ahmed Bassiouny, Assisstant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12020
Record Dates: First submitted 2020-04-18; First posted 2020-04-22 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Intervention Model Description: Two groups of poor ovarian responders to be given two different induction protocols at the same time duration of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimal Stimulation Group (Active Comparator): Minimal dose stimulation ovarian induction protocol given to poor responders, involving letrozole, low dose recombinant FSH and GnRH antagonist
  Interventions: Drug: Minimal stimulation protocol; Procedure: IVF/ICSI cycle
- Microflare Group (Active Comparator): Microflare ovarian induction protocol given to poor responders, involving OCP, GnRH agonist, high dose recombinant FSH
  Interventions: Drug: Microflare protocol; Procedure: IVF/ICSI cycle

INTERVENTIONS:
Drug: Minimal stimulation protocol — Letrozole, Recombinant FSH, GnRH antagonist
  Other Names: Ovarian induction protocol
  Arms: Minimal Stimulation Group
Drug: Microflare protocol — OCP, GnRH agonist, Recombinant FSH
  Other Names: Ovarian induction protocol
  Arms: Microflare Group
Procedure: IVF/ICSI cycle — Involving ovum pickup and embryo transfer

SUMMARY:
Comparing two ovarian induction protocols in poor responders in IVF/ICSI cycles

DETAILED DESCRIPTION:
The two groups of poor responders are randomized into either; a minimal dose stimulation protocol involving letrozole, recombinant FSH and GnRH antagonist versus a microflare conventional protocol with OCP, GnRH agonist and high dose recombinant FSH, in their IVF/ICSI cycles, primary outcome will be the number of oocytes retrieved.

ELIGIBILITY:
Inclusion Criteria:

1- More than 1 year of infertility 2 - Poor ovarian responder according to the Bologna criteria:

1. Advanced maternal age
2. Previous poor ovarian response
3. Abnormal tests of ovarian reserve (AFC < 5-7, AMH <0.5-1.1 ng/ml)

Exclusion Criteria:

1. Age > 43 years
2. baseline FSH >15 mIU/ml
3. Previous ovarian surgery
4. Ovarian endometrioma
5. Uterine anomaly or myoma
6. Any medical disorder
7. Any hormonal disorder eg. hyperprolactinemia
8. BMI > 30 kg/m2
9. Severe male factor

Ages: 30 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Number of oocytes retrieved | 10 to 14 days
  the number of oocytes collected from each participants in the two groups on the day of ovum pickup

SECONDARY OUTCOMES:
Number of MII oocytes retrieved | 10 to 14 days
  The mature oocytes colloected on the day of ovum pickup
Number of fertilized oocytes | 2 days
  Number of oocytes fertilized
Number of embryos transferred | Day 3 after ovum pickup
  Number of embryos transferred in the induction cycle
Number of embryos cryopreserved | Day 3 after ovum pickup
  Any surplus good quality embryos available for cryopreservation
Chemical pregnancy rate | 14 days after embryo ransfer
  Positive pregnancy test
Clinical pregnancy rate | 5 to 7 weeks after embryo transfer
  Positive heart beat
Early miscarriage rate | 12 weeks
  loss of pregnancy before 12 weeks
Ongoing pregnancy rate | 12 weeks
  pregnancy beyond 12 weeks
Live birth rate | 28 to 40 weeks
  Delivery beyond 28 weeks

OTHER OUTCOMES:
Cancellation rate | 10 to 14 days
  Number of cycles not reaching ovum pickup
Total dose of recombinant FSH | 10 to 14 days
  The mean total dose of recombinant FSH used in the cycle of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sarwat Ahwany, MD, Study Director — Cairo University
Locations (2):
- Egypt (2):
  - IVF centre, Obstetrics and Gynaecology Department, Cairo University Hospitals (Kasr EL Aini), Cairo
  - Cairo University, Cairo